CLINICAL TRIAL: NCT02509208
Title: A Multicenter Study to Assess the Safety and Performance of SurgiClot® in the Treatment of Cancellous Bone Bleeding
Brief Title: A Study to Assess the Safety and Performance of SurgiClot® in the Treatment of Cancellous Bone Bleeding
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Teresa Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STM-UK-001
Record Dates: First submitted 2015-07-22; First posted 2015-07-27 (Estimated); Last update posted 2017-04-27 (Actual); Status verified 2017-04

CONDITIONS: Cancellous Bone Bleeding
Keywords: iliac crest bone graft; ICBG; pelvic osteotomy; spinal fusion; hemostasis; haemostasis; hemostatic; haemostatic; dextran; SurgiClot; cancellous bone bleeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SurgiClot (Experimental): All qualified subjects will be treated with the SurgiClot haemostatic dressing
  Interventions: Device: SurgiClot haemostatic dressing

INTERVENTIONS:
Device: SurgiClot haemostatic dressing — haemostatic dressing

SUMMARY:
The purpose of this European study is to demonstrate the safety and performance of the SurgiClot® dressing in the treatment of cancellous bone bleeding.

DETAILED DESCRIPTION:
Patients who require surgery for iliac crest bone graft (ICBG), pelvic osteotomy or spinal fusion will be screened for this multicenter, prospective, non-randomized, open-label study. All qualified subjects will be treated with the SurgiClot® haemostatic dressing (a completely soluble dressing consisting of solid nanofibers of electrospun dextran with embedded lyophilized human fibrinogen and thrombin proteins).

The safety and performance of the SurgiClot dressing will be evaluated in up to 40 subjects enrolled in Europe. Subjects will be followed for six weeks after the surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing a planned elective orthopaedic or spinal surgical procedure. Spinal surgery can be the entire spine although it should be confined to one or two-level fusions e.g. one or two level cervical, or thoracic or lumbar.
* Patient has an intraoperative bleeding site involving cancellous bone that the surgeon would typically treat with another topical haemostatic agent to control the bleeding.
* Patient has normal liver function
* The subject is willing and able to comply with the requirements of the study protocol, including the six weeks follow-up evaluation.

Exclusion Criteria:

* Is unable or unwilling to return for the follow-up visit.
* The subject has had surgery at the intended application site ≤ 6 months before the current surgical procedure.
* Active infection at the surgical site.
* Pregnancy, as determined by urine pregnancy test, or breast feeding.
* Pre-operative platelet count < 150,000, INR > 1.3, and/or APTT > 32.4.
* Pre-operative anaemia (Hb < 110 g/L in females, Hb < 120 g/L in males).
* Use of anticoagulant therapy (e.g., coumadin, heparin, clopidogrel), non-steroidal anti-inflammatory medications or fish oil supplements within 7 days of the surgery except for aspirin. (maximum dose 150 mg per day)
* Patient with a blood dyscrasia.
* Presence of a spinal tumour, intradural pathology, or prior spinal fusion surgery at the same target site.
* Participation in another clinical trial with an investigational drug or device within the past 30 days.
* Known allergy to human fibrinogen, human thrombin, or porcine-derived products.
* Compromised immune system.
* The use of a haemostatic agent is contraindicated for the subject.
* Fibrinolytic disorders requiring intraoperative antifibrinolytic treatment.
* Haematological disease (thromboembolic events, haemoglobinopathy, coagulopathy or haemolytic disease)
* Significant co-morbidities: Previous myocardial infarction (MI); severe ischemic heart disease (New York Heart Association Class III, IV); severe pulmonary disease; chronic renal failure; hepatic failure; uncontrolled hypertension.
* Subject is unwilling to receive blood products.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-07; Primary Completion 2016-01 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
The proportion of patients that achieve controlled haemostasis at the target bleeding site at 3 minutes | 3 minutes
Incidence of device-related adverse events | 6 weeks

SECONDARY OUTCOMES:
Proportion of patients needing a repeat application of the dressing | intra-operative
Proportion of repeat applications that achieve haemostasis | intra-operative
Proportion of patients with negative immunogenicity response of coagulation factors: prothrombin time (PT) | 6 weeks
Proportion of patients with negative immunogenicity response of coagulation factors: activated partial thromboplastin time (aPTT) | 6 weeks
Proportion of patients with negative immunogenicity response of coagulation factors: international normalized ratio (INR) | 6 weeks
Proportion of patients with negative immunogenicity response of coagulation factors: fibrinogen | 6 weeks
Assess dressing characteristics of dissolvability via scales on a Product-Handling Characteristics Questionnaire | intra-operative
Assess dressing characteristics of ease of preparation via scales on a Product-Handling Characteristics Questionnaire | intra-operative
Assess dressing characteristics of conformability via scales on a Product-Handling Characteristics Questionnaire | intra-operative
Assess dressing characteristics of ease of use via scales on a Product-Handling Characteristics Questionnaire | intra-operative
Mean volume of blood loss through the standard of care of the hospital | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Niall Craig, MD, Principal Investigator — Aberdeen Royal Infirmary
Locations (8):
- Norway (2):
  - Helse Møre og Romsdal HF, Ålesund sjukehus, Ålesund
  - Helse Møre og Romsdal HF, Kristiansund sjukehus, Kristiansund
- United Kingdom (6):
  - Salford Royal Infirmary, Salford, Manchester
  - Jones & Hunt Orthopaedic Hospital, Oswestry, Shropshire
  - Doncaster Royal Infirmary, Doncaster, Yorkshire
  - Aberdeen Royal Infirmary, Aberdeen
  - Castle Hill Hospital, Cottingham
  - Royal Victoria Infirmary, Newcastle upon Tyne